CLINICAL TRIAL: NCT04689750
Title: Impact of Donor Clonal Haematopoiesis of Indeterminate Potential (CHIP) on Recipient Outcome Following Allogeneic Haematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: Donor CHIP and Allogeneic HSCT Outcome
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: CHIP001
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Clonal Hematopoiesis
Keywords: Donor clonal hematopoiesis; Allogeneic hematopoiectic stem cell transplantation; Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood or bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic HSCT recipients and donors
  Interventions: Diagnostic Test: Next generation sequencing

INTERVENTIONS:
Diagnostic Test: Next generation sequencing — Genetic profile of donors will be collected at the time of PBSC or BM stem cell donation. Genetic profile of recipients will be collected at 1-month, 6-month, 12-month post-HSCT and at time of relapse or occurrence of leukaemia.
  Gene mutations and pathogenic gene fusion will be determined in the peripheral blood and/or marrow samples by next-generation sequencing (NGS) using a myeloid-gene panel and nanopore long-read sequencing.

SUMMARY:
Current data on the impact of donor CHIP on long-term recipient outcome remain largely speculative. Data on the impact of donor CHIP including on allograft function, immunologic dysfunction, graft versus host disease (GVHD), disease relapse and survival across various donor populations are scarce. This is a retrospective-prospective cohort study designed to determine the association between donor gene mutations and outcome following allogeneic HSCT.

DETAILED DESCRIPTION:
This is a single centre prospective and retrospective cohort study. This study involves allo-HSCT recipients and their donors at Queen Mary Hospital, Hong Kong. Information on the presence of gene mutations in donor peripheral blood or bone marrow sample; gene mutations in recipient peripheral blood or bone marrow post-allo-HSCT; and donor and recipient outcome will be collected in either prospective, partial-prospective/retrospective or retrospective manner. The information will be used to determine the association between the presence of clonal haematopoiesis in the donor and recipient outcome following allo-HSCT.

Data will be collected through routine clinical visits and/or reviewing medical records. Data will be collected at the time of peripheral blood stem cells (PBSC) or bone marrow stem cells donation, at the time of allo-HSCT, one month post-allo-HSCT and every 6 months thereafter until death/study termination.

Genetic profile of donors will be collected at the time of PBSC or BM stem cell donation. Genetic profile of recipients will be collected at 1-month, 6-month, 12-month post-HSCT and at time of relapse or occurrence of leukaemia.

Gene mutations and pathogenic gene fusion will be determined in the peripheral blood and/or marrow samples by next-generation sequencing (NGS) using a myeloid-gene panel and nanopore long-read sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 year or above
2. Donor and recipient of allo-HSCT
3. In prospective and partial prospective/retrospective case, subjects who have provided a signed written informed consent. In retrospective case, subjects who had provided a previously signed written informed consent on:

   1. voluntary provision of clinical data, and
   2. voluntary provision of archived/remaining specimens for genetic analysis, and
   3. authorizing storage and usage of archived/remaining specimens for any further analysis

Exclusion Criteria:

1. Autologous peripheral blood stem cells or bone marrow stem cell donors for autologous HSCT

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve allo-HSCT recipients and their donors at Queen Mary Hospital, Hong Kong. Information on the presence of gene mutations in donor peripheral blood or bone marrow sample; gene mutations in recipient peripheral blood or bone marrow post-allo-HSCT; and donor and recipient outcome will be collected in either prospective, partial-prospective/retrospective or retrospective manner.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) of the recipient. | 5 years
  This is defined as the time (in months) from the date of allo-HSCT to death from any cause (event), latest follow-up (censor) or study termination.
Progression-free survival (PFS) of the recipient. | 5 years
  This is defined as the time (in months) from the date of allo-HSCT to relapse/progression (event), death, latest follow-up or study termination.

SECONDARY OUTCOMES:
Acute and chronic GVHD | 5 years
  The occurrence of acute and/or chronic graft-versus-host disease
Leukemia of donor origin | 5 years
  The occurrence of donor cell derived MDS/AML in the recipient following allogeneic HSCT
Cardiac complications | 5 years
  The occurrence of arrthymias, pericardial disease, coronary artery disease, myocardial dysfunction, pulmonary hypertension
Pulmonary complications | 5 years
  The occurrence of bronchiolitis obliterans, bronchiolitis obliterans with organizing pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steensma DP, Bejar R, Jaiswal S, Lindsley RC, Sekeres MA, Hasserjian RP, Ebert BL. Clonal hematopoiesis of indeterminate potential and its distinction from myelodysplastic syndromes. Blood. 2015 Jul 2;126(1):9-16. doi: 10.1182/blood-2015-03-631747. Epub 2015 Apr 30. PMID 25931582
- [Background] Steensma DP, Ebert BL. Clonal hematopoiesis as a model for premalignant changes during aging. Exp Hematol. 2020 Mar;83:48-56. doi: 10.1016/j.exphem.2019.12.001. Epub 2019 Dec 12. PMID 31838005
- [Background] Steensma DP. Clinical Implications of Clonal Hematopoiesis. Mayo Clin Proc. 2018 Aug;93(8):1122-1130. doi: 10.1016/j.mayocp.2018.04.002. Epub 2018 Jul 4. PMID 30078412
- [Background] Steensma DP. Clinical consequences of clonal hematopoiesis of indeterminate potential. Blood Adv. 2018 Nov 27;2(22):3404-3410. doi: 10.1182/bloodadvances.2018020222. PMID 30482770
- [Background] Shlush LI, Zandi S, Mitchell A, Chen WC, Brandwein JM, Gupta V, Kennedy JA, Schimmer AD, Schuh AC, Yee KW, McLeod JL, Doedens M, Medeiros JJ, Marke R, Kim HJ, Lee K, McPherson JD, Hudson TJ; HALT Pan-Leukemia Gene Panel Consortium; Brown AM, Yousif F, Trinh QM, Stein LD, Minden MD, Wang JC, Dick JE. Identification of pre-leukaemic haematopoietic stem cells in acute leukaemia. Nature. 2014 Feb 20;506(7488):328-33. doi: 10.1038/nature13038. Epub 2014 Feb 12. PMID 24522528
- [Background] Gibson CJ, Kennedy JA, Nikiforow S, Kuo FC, Alyea EP, Ho V, Ritz J, Soiffer R, Antin JH, Lindsley RC. Donor-engrafted CHIP is common among stem cell transplant recipients with unexplained cytopenias. Blood. 2017 Jul 6;130(1):91-94. doi: 10.1182/blood-2017-01-764951. Epub 2017 Apr 26. PMID 28446434
- [Background] Frick M, Chan W, Arends CM, Hablesreiter R, Halik A, Heuser M, Michonneau D, Blau O, Hoyer K, Christen F, Galan-Sousa J, Noerenberg D, Wais V, Stadler M, Yoshida K, Schetelig J, Schuler E, Thol F, Clappier E, Christopeit M, Ayuk F, Bornhauser M, Blau IW, Ogawa S, Zemojtel T, Gerbitz A, Wagner EM, Spriewald BM, Schrezenmeier H, Kuchenbauer F, Kobbe G, Wiesneth M, Koldehoff M, Socie G, Kroeger N, Bullinger L, Thiede C, Damm F. Role of Donor Clonal Hematopoiesis in Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2019 Feb 10;37(5):375-385. doi: 10.1200/JCO.2018.79.2184. Epub 2018 Nov 7. PMID 30403573
- [Background] Wong WH, Bhatt S, Trinkaus K, Pusic I, Elliott K, Mahajan N, Wan F, Switzer GE, Confer DL, DiPersio J, Pulsipher MA, Shah NN, Sees J, Bystry A, Blundell JR, Shaw BE, Druley TE. Engraftment of rare, pathogenic donor hematopoietic mutations in unrelated hematopoietic stem cell transplantation. Sci Transl Med. 2020 Jan 15;12(526):eaax6249. doi: 10.1126/scitranslmed.aax6249. PMID 31941826